CLINICAL TRIAL: NCT05929027
Title: Self-Administered Gaming and Exercise at Home (SAGEH)
Acronym: SAGEH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Sheikh Khalifa Stroke Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00340964
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Stroke; Hand Weakness
Keywords: stroke; stroke recovery; hand weakness; video game
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Arm G1 (Active Comparator): The interventions will consist of 5 daily sessions over 3 weeks. Because the interventions are self-administered, the sessions are unsupervised in the sense that the sessions do not include synchronous therapy provided by a clinician or a therapist. Instead, during each week, the intervention will include 2 short (less than 15 minutes) telemedicine check-in appointments (not standard of care) provided by a licensed occupational therapist for the purposes of assessing safety and providing guidance for the unsupervised sessions. The intervention will focus on stretches, warm-up and strengthening exercises aimed at improving hand function.
  Interventions: Behavioral: occupational therapy - self directed
- Treatment Arm G2 (Experimental): The intervention will consist of 5 daily sessions over 3 weeks. Because the interventions are self-administered, the sessions are unsupervised in the sense that the sessions do not include synchronous therapy provided by a clinician or a therapist. Instead, during each week, the intervention will include 2 short (less than 15 minutes) telemedicine check-in appointments (not standard of care) provided by a licensed occupational therapist for the purposes of assessing safety and providing guidance for the unsupervised sessions. In this treatment arm, participants will use a knob-like computer interface connected to a tablet. The tablet features a series of game-like tasks to be carried out by moving the interface with the fingers. The target intervention is scheduled for 1.5 hours per day, which is typically divided into two sessions of 40 minutes with a 10-minute break in between.
  Interventions: Behavioral: NoNo
- Control Group (CG) (No Intervention): Unlike G1 and G2, the CG will remain in the standard of care treatment plan but will not receive any additional therapy. That is to say, participants will follow standard therapy plans as dictated by normal post-stroke hospital discharge planning. The only difference from the standard of care will be that participants in CG will still receive identical check-in appointments with follow-up questions concerning recovery and activities.

INTERVENTIONS:
Behavioral: NoNo — Participants in the G2 group will use the Twirlstone (knob-like) device to play a videogame called Nono's World. The Twirlstone is an electromechanical device that resembles a knob and a standard joystick (identical to the discontinued Atari CX-20 Controller). The knob can rotate or move in a push-pull fashion. To control the game's character (an axolotl called Nono), a signal about the knob motion is relayed to the computer wirelessly. This device has been certified by Johns Hopkins University's Clinical Engineering Services, where it was deemed less than minimum risk. The game has been custom built to allow participants to take control of the character using subtle manipulative finger movements to accomplish game-like tasks.
  The investigators will use portable communication devices to carry out telemedicine sessions. All devices and are low-power battery-operated tools for encouraging hand movement and the components are approved for use in the commercial market.
  Arms: Treatment Arm G2
Behavioral: occupational therapy - self directed — Participants 5 daily sessions over 3 weeks consisting of self-administered, unsupervised occupational therpay. Additionally, participants will have 2, <15 minutes telemedicine check-in appointments (not standard of care) provided by a licensed occupational therapist for the purposes of assessing safety and providing guidance for the unsupervised sessions. The intervention will focus on stretches, warm-up and strengthening exercises aimed at improving hand function.
  The investigators will use portable communication devices for the purposes of carrying out telemedicine sessions. All devices and are low-power battery-operated tools for encouraging hand movement and the components are approved for use in the commercial market.
  Arms: Treatment Arm G1

SUMMARY:
This study aims at comparing manual function outcomes between the standard of care and additional self-administered hand therapy after stroke. Strokes are common neurological injuries, and although rates of survival have increased in recent decades, survivors often continue to experience deficiencies in hand dexterity and bimanual function. Most motor recovery takes place within the first 3 months after a stroke. This initial period is necessary for stabilizing the patient but also provides different opportunities to foster motor recovery. Functional gains, including instances after the post-acute period, have been observed after regular and frequent (high dosage) therapy, suggesting that recovery is likely influenced by practice-driven sensorimotor learning. These findings motivate the implementation of daily therapeutic regimes beyond post-stroke hospitalization and basic motor function, aiming instead at addressing overlooked deficiencies in manipulation and bimanual coordination. While some hand therapy is often provided during outpatient therapy visits (the standard of care), self-administered sessions play a large role in implementing additional daily therapy. As a result, the investigators are interested in both the implementation of self-administered regimes and measuring clinical outcomes with and without self-administered therapy.

DETAILED DESCRIPTION:
The primary goal of this study is to determine if adding self-administered, daily hand therapy to standard of care improves post-stroke clinical outcomes. The investigators will investigate two distinct approaches to implement self-administered therapy and observe how the participants fare to the standard outpatient visits-a total of 3 experimental groups. The first approach consists of daily exercise routines; the second approach consists of using a novel, portable, electronic device that was intentionally designed to address the difficult problem of hand rehabilitation. Specifically, the device combines hand therapy with video game-like tasks. Both post-stroke approaches will be partially supervised by an occupational therapist via short telemedicine sessions, in the context of standard-of-care telemedicine clinic (JSTTEP - described below) to promote safety and proper form during the exercises or device utilization.

The primary outcome is a standardized, post-intervention functional hand metric. This pilot study will include both measurement of improvements with respect to a baseline, and comparison between groups, using the therapist-provided therapy sessions as control and gold standard.

The investigators will recruit 60 adult stroke survivors. The total will be divided into three matched groups. Two of the groups (G1 and G2, 20 participants each) will receive therapy-based interventions in addition to the standard of care, and the remaining control group (CG, 20 participants) will receive the standard of care and no additional therapy.

Current standard of care regarding stroke inpatients requires admission to Johns Hopkins Comprehensive Stroke Center. At discharge, depending upon the stroke severity, patients can either be discharged to a facility or to home. This study is specifically targeting patients discharged to home.

Importantly, patients going home are followed in the Joint Stroke Transitional Technology-Enhanced Program (JSTTEP). JSTTEP is the standard of care, inter-disciplinary, telemedicine program that operates during the first month after stroke to facilitate the patient's transition from hospital to home. Each shared visit includes a physician and therapist evaluation and combined treatment plan. A single multidisciplinary online group education session is completed within 1 month after stoke hospitalization and is open to patients and care partners.

Stroke patients who are being discharged home from the Johns Hopkins Comprehensive Stroke Center via JSTTEP are eligible for participation in this study. A consecutive series of patients who meet inclusion criteria will be approached for consent to participate in this study. Inclusion (or exclusion) will be determined using the criteria described in the Inclusion/Exclusion Criteria Section, using a HIPAA Privacy Authorization Form. Upon consenting to participate in the study, each participant will undergo a Baseline Assessment visit, while still an inpatient, composed of a gaming, functional, and cognitive assessments (described below under Baseline Assessment). These assessments also work as screenings; that is, if, after signing the consent and during the enrollment process, a patient fails to meet enrollment criteria, the investigators can halt enrollment. Similarly, if a patient does meet the enrollment criteria, the participants will be assigned into a treatment group (as described below in the Randomization Section), and will receive instructions according to the participants group

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years and over
2. Stroke confirmed by CT or MRI within the previous 6 weeks.
3. Arm and/or hand impairment induced by the stroke.
4. Meet JSTTEP criteria and are enrolled in JSTTEP.
5. Admitted to the Johns Hopkins Hospital (JHH) inpatient stroke service.
6. Proficient in speaking and reading English.
7. Willing and capable to contacted remotely for all necessary telemedicine contacts.
8. No history of prior ischemic or hemorrhagic stroke with associated motor deficits (prior stroke with no upper limb motor symptoms is allowed)
9. Ability to give informed consent.

Exclusion Criteria:

1. Arm impairment that is too severe (FM-UE < 40) on day of baseline testing prior to beginning of the study.
2. Recent Botox injection to upper limb (since stroke onset).
3. History of physical or neurological condition that interferes with study procedures or assessment of motor function (e.g. severe arthritis, severe neuropathy, Parkinson's disease).
4. Terminal illness with life expectancy < 6 months.
5. Inability to sit in a chair and perform hand exercises for 20 minutes at the time.
6. Cognitive impairment, with score on Montreal Cognitive Assessment (MoCA) ≤ 20.
7. Social and/or personal circumstances that prevent telemedicine follow-up.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in finger dexterity as assessed by the nine-hole peg test (9PHT) | Baseline, post-intervention up to 7 days, 6 months post-stroke
  The Nine-Hole Peg Test (9HPT) is used to measure finger dexterity in patients with various neurological diagnoses. Participants are asked to place pegs into the holes one at a time, then remove them one at a time, and place them back in the container as fast as they can.

SECONDARY OUTCOMES:
Change in arm hand function using the Fugl Meyer Scale. | Baseline, up to 7 days post-intervention, and 6 months post-stroke
  Change in arm and hand function at the impairment level as assessed by the Fugl Meyer Upper Extremity Assessment of motor control (FM-UE). The FM-UE uses a 3-point ordinal scale to evaluate sensorimotor function of the arm and hand of the affected upper extremity during reach and grasp movements in and out of synergistic movement patterns
Change in arm and hand function using the ARAT | Baseline, up to 7 days post-intervention, and 6 months post-stroke
  Change in arm and hand function at the activity level as assessed by the Action Research Arm Test (ARAT). The ARAT is a 19-item measure with 4 subtests (grip, grasp, pinch, and gross arm movement) and 57 possible points. Each subtest has tasks varying in complexity that are graded using a 4-point ordinal scale to describe if tasks are completed with normal movement, movement that requires increased time, are partially completed, or unable to be completed.
Change in fingertip individuation index as assessed by the Cyber Glove | Baseline, up to 7 days post-intervention, and 6 months post-stroke
  Change in fingertip individuation index as assessed by kinematic measurement of digit movement using the CyberGlove. The Cyberglove is a wearable device that uses sensor-based technology to capture joint range of motion. Full extension and flexion of each digit in isolation will be captured using this technology.
Change in Cognitive impairment as assessed by Montreal Cognitive Assessment (MOCA) | Baseline, up to 7 days post-intervention, and 6 months post-stroke
  Montreal Cognitive Assessment (MOCA) will be used. The MOCA is a screening assessment for mild cognitive impairment. It has 30 questions that assess different domains of cognition including: executive functions, memory, language, attention, and abstract reasoning.
Engagement and enjoyment of the different sub-aspects within each additional therapy approach as assessed by satisfaction surveys developed by the study team | up to 7 days post--intervention
  Engagement and enjoyment of the different sub-aspects within each additional therapy approach as assessed by satisfaction surveys which will contain a combination of questions including Likert scale-based questions, ordinal questions, and fill-in-the-blank questions (the study team will create this survey specific for this study.
Change in disability as assessed by the modified Rankin score | Baseline, up to 7 days pot-intervention, and 6 months post-stroke
  Change in disability as assessed by the modified Rankin Scale (mRS). The mRS is a widely used clinician reported , single-item measure of global disability

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Zeiler, M.D, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkin, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johansson GM, Hager CK. A modified standardized nine hole peg test for valid and reliable kinematic assessment of dexterity post-stroke. J Neuroeng Rehabil. 2019 Jan 14;16(1):8. doi: 10.1186/s12984-019-0479-y. PMID 30642350
- [Background] Bejot Y, Daubail B, Giroud M. Epidemiology of stroke and transient ischemic attacks: Current knowledge and perspectives. Rev Neurol (Paris). 2016 Jan;172(1):59-68. doi: 10.1016/j.neurol.2015.07.013. Epub 2015 Dec 21. PMID 26718592
- [Background] Heron M. Deaths: Leading Causes for 2019. Natl Vital Stat Rep. 2021 Jul;70(9):1-114. PMID 34520342
- [Background] Brunnstrom S. Motor testing procedures in hemiplegia: based on sequential recovery stages. Phys Ther. 1966 Apr;46(4):357-75. doi: 10.1093/ptj/46.4.357. No abstract available. PMID 5907254
- [Background] Nakayama H, Jorgensen HS, Raaschou HO, Olsen TS. Recovery of upper extremity function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1994 Apr;75(4):394-8. doi: 10.1016/0003-9993(94)90161-9. PMID 8172497
- [Background] Kotila M, Waltimo O, Niemi ML, Laaksonen R, Lempinen M. The profile of recovery from stroke and factors influencing outcome. Stroke. 1984 Nov-Dec;15(6):1039-44. doi: 10.1161/01.str.15.6.1039. PMID 6506115
- [Background] Colebatch JG, Gandevia SC. The distribution of muscular weakness in upper motor neuron lesions affecting the arm. Brain. 1989 Jun;112 ( Pt 3):749-63. doi: 10.1093/brain/112.3.749. PMID 2731028
- [Background] Jebsen RH, Taylor N, Trieschmann RB, Trotter MJ, Howard LA. An objective and standardized test of hand function. Arch Phys Med Rehabil. 1969 Jun;50(6):311-9. No abstract available. PMID 5788487
- [Background] Barry AJ, Triandafilou KM, Stoykov ME, Bansal N, Roth EJ, Kamper DG. Survivors of Chronic Stroke Experience Continued Impairment of Dexterity But Not Strength in the Nonparetic Upper Limb. Arch Phys Med Rehabil. 2020 Jul;101(7):1170-1175. doi: 10.1016/j.apmr.2020.01.018. Epub 2020 Feb 28. PMID 32113974
- [Background] Krakauer JW, Kitago T, Goldsmith J, Ahmad O, Roy P, Stein J, Bishop L, Casey K, Valladares B, Harran MD, Cortes JC, Forrence A, Xu J, DeLuzio S, Held JP, Schwarz A, Steiner L, Widmer M, Jordan K, Ludwig D, Moore M, Barbera M, Vora I, Stockley R, Celnik P, Zeiler S, Branscheidt M, Kwakkel G, Luft AR. Comparing a Novel Neuroanimation Experience to Conventional Therapy for High-Dose Intensive Upper-Limb Training in Subacute Stroke: The SMARTS2 Randomized Trial. Neurorehabil Neural Repair. 2021 May;35(5):393-405. doi: 10.1177/15459683211000730. Epub 2021 Mar 20. PMID 33745372
- [Background] Murphy TH, Corbett D. Plasticity during stroke recovery: from synapse to behaviour. Nat Rev Neurosci. 2009 Dec;10(12):861-72. doi: 10.1038/nrn2735. Epub 2009 Nov 4. PMID 19888284
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] BENNETT EL, DIAMOND MC, KRECH D, ROSENZWEIG MR. CHEMICAL AND ANATOMICAL PLASTICITY BRAIN. Science. 1964 Oct 30;146(3644):610-9. doi: 10.1126/science.146.3644.610. No abstract available. PMID 14191699
- [Background] McDonald MW, Hayward KS, Rosbergen ICM, Jeffers MS, Corbett D. Is Environmental Enrichment Ready for Clinical Application in Human Post-stroke Rehabilitation? Front Behav Neurosci. 2018 Jul 11;12:135. doi: 10.3389/fnbeh.2018.00135. eCollection 2018. PMID 30050416
- [Background] Vive S, Af Geijerstam JL, Kuhn HG, Bunketorp-Kall L. Enriched, Task-Specific Therapy in the Chronic Phase After Stroke: An Exploratory Study. J Neurol Phys Ther. 2020 Apr;44(2):145-155. doi: 10.1097/NPT.0000000000000309. PMID 32118616
- [Background] Platz T. Impairment-oriented training (IOT)--scientific concept and evidence-based treatment strategies. Restor Neurol Neurosci. 2004;22(3-5):301-15. PMID 15502273
- [Background] Platz T, Lotze M. Arm Ability Training (AAT) Promotes Dexterity Recovery After a Stroke-a Review of Its Design, Clinical Effectiveness, and the Neurobiology of the Actions. Front Neurol. 2018 Dec 11;9:1082. doi: 10.3389/fneur.2018.01082. eCollection 2018. PMID 30619042
- [Background] Krakauer JW, Cortes JC. A non-task-oriented approach based on high-dose playful movement exploration for rehabilitation of the upper limb early after stroke: A proposal. NeuroRehabilitation. 2018;43(1):31-40. doi: 10.3233/NRE-172411. PMID 30056438
- [Background] Schieber MH, Santello M. Hand function: peripheral and central constraints on performance. J Appl Physiol (1985). 2004 Jun;96(6):2293-300. doi: 10.1152/japplphysiol.01063.2003. PMID 15133016
- [Background] Elliott JM, Connolly KJ. A classification of manipulative hand movements. Dev Med Child Neurol. 1984 Jun;26(3):283-96. doi: 10.1111/j.1469-8749.1984.tb04445.x. PMID 6734945
- [Background] Xu J, Ejaz N, Hertler B, Branscheidt M, Widmer M, Faria AV, Harran MD, Cortes JC, Kim N, Celnik PA, Kitago T, Luft AR, Krakauer JW, Diedrichsen J. Separable systems for recovery of finger strength and control after stroke. J Neurophysiol. 2017 Aug 1;118(2):1151-1163. doi: 10.1152/jn.00123.2017. Epub 2017 May 31. PMID 28566461
- [Background] Raghavan P, Santello M, Gordon AM, Krakauer JW. Compensatory motor control after stroke: an alternative joint strategy for object-dependent shaping of hand posture. J Neurophysiol. 2010 Jun;103(6):3034-43. doi: 10.1152/jn.00936.2009. Epub 2010 Mar 24. PMID 20457866
- [Background] Patel P, Kaingade SR, Wilcox A, Lodha N. Force control predicts fine motor dexterity in high-functioning stroke survivors. Neurosci Lett. 2020 Jun 11;729:135015. doi: 10.1016/j.neulet.2020.135015. Epub 2020 Apr 30. PMID 32360934
- [Background] Karni A, Meyer G, Rey-Hipolito C, Jezzard P, Adams MM, Turner R, Ungerleider LG. The acquisition of skilled motor performance: fast and slow experience-driven changes in primary motor cortex. Proc Natl Acad Sci U S A. 1998 Feb 3;95(3):861-8. doi: 10.1073/pnas.95.3.861. PMID 9448252
- [Background] Cramer SC, Dodakian L, Le V, See J, Augsburger R, McKenzie A, Zhou RJ, Chiu NL, Heckhausen J, Cassidy JM, Scacchi W, Smith MT, Barrett AM, Knutson J, Edwards D, Putrino D, Agrawal K, Ngo K, Roth EJ, Tirschwell DL, Woodbury ML, Zafonte R, Zhao W, Spilker J, Wolf SL, Broderick JP, Janis S; National Institutes of Health StrokeNet Telerehab Investigators. Efficacy of Home-Based Telerehabilitation vs In-Clinic Therapy for Adults After Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Sep 1;76(9):1079-1087. doi: 10.1001/jamaneurol.2019.1604. PMID 31233135
- [Background] Raglio A, Panigazzi M, Colombo R, Tramontano M, Iosa M, Mastrogiacomo S, Baiardi P, Molteni D, Baldissarro E, Imbriani C, Imarisio C, Eretti L, Hamedani M, Pistarini C, Imbriani M, Mancardi GL, Caltagirone C. Hand rehabilitation with sonification techniques in the subacute stage of stroke. Sci Rep. 2021 Mar 31;11(1):7237. doi: 10.1038/s41598-021-86627-y. PMID 33790343
- [Background] Unibaso-Markaida I, Iraurgi I, Ortiz-Marques N, Amayra I, Martinez-Rodriguez S. Effect of the Wii Sports Resort on the improvement in attention, processing speed and working memory in moderate stroke. J Neuroeng Rehabil. 2019 Feb 28;16(1):32. doi: 10.1186/s12984-019-0500-5. PMID 30819204
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Tariq SH, Tumosa N, Chibnall JT, Perry MH 3rd, Morley JE. Comparison of the Saint Louis University mental status examination and the mini-mental state examination for detecting dementia and mild neurocognitive disorder--a pilot study. Am J Geriatr Psychiatry. 2006 Nov;14(11):900-10. doi: 10.1097/01.JGP.0000221510.33817.86. PMID 17068312
- [Background] Reuben DB, Magasi S, McCreath HE, Bohannon RW, Wang YC, Bubela DJ, Rymer WZ, Beaumont J, Rine RM, Lai JS, Gershon RC. Motor assessment using the NIH Toolbox. Neurology. 2013 Mar 12;80(11 Suppl 3):S65-75. doi: 10.1212/WNL.0b013e3182872e01. PMID 23479547
- [Background] Wilson PH, Rogers JM, Vogel K, Steenbergen B, McGuckian TB, Duckworth J. Home-based (virtual) rehabilitation improves motor and cognitive function for stroke patients: a randomized controlled trial of the Elements (EDNA-22) system. J Neuroeng Rehabil. 2021 Nov 25;18(1):165. doi: 10.1186/s12984-021-00956-7. PMID 34823545
- [Background] Beebe JA, Lang CE. Relationships and responsiveness of six upper extremity function tests during the first six months of recovery after stroke. J Neurol Phys Ther. 2009 Jun;33(2):96-103. doi: 10.1097/NPT.0b013e3181a33638. PMID 19556918
- [Background] Schneider EJ, Ada L, Lannin NA. Extra upper limb practice after stroke: a feasibility study. Pilot Feasibility Stud. 2019 Dec 30;5:156. doi: 10.1186/s40814-019-0531-5. eCollection 2019. PMID 31893129
- [Background] Heshmatollah A, Dommershuijsen LJ, Fani L, Koudstaal PJ, Ikram MA, Ikram MK. Long-term trajectories of decline in cognition and daily functioning before and after stroke. J Neurol Neurosurg Psychiatry. 2021 Nov;92(11):1158-1163. doi: 10.1136/jnnp-2021-326043. Epub 2021 Jul 6. PMID 34230107
- [Background] Heller A, Wade DT, Wood VA, Sunderland A, Hewer RL, Ward E. Arm function after stroke: measurement and recovery over the first three months. J Neurol Neurosurg Psychiatry. 1987 Jun;50(6):714-9. doi: 10.1136/jnnp.50.6.714. PMID 3612152